CLINICAL TRIAL: NCT00972062
Title: Herbal Therapy for Subcutaneous Injection Site Reactions in Multiple Sclerosis
Acronym: MSSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TEVA 540837
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis
Keywords: Subcutaneous injections; Skin abnormalities
MeSH Terms: conditions — Multiple Sclerosis; Skin Abnormalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo cream (Placebo Comparator): Cream base used in compounding medications into cream media
  Interventions: Other: Placebo Cream
- Herbal Cream (Experimental): Herbal cream (Bach's Rescue Remedy Cream) applied to skin site reactions from MS medications
  Interventions: Other: Bach's Rescue Remedy Cream

INTERVENTIONS:
Other: Bach's Rescue Remedy Cream — 0.5 ml of cream applied to skin site reactions as needed
  Other Names: Rescue Cream
  Arms: Herbal Cream
Other: Placebo Cream — Placebo cream 0.5 ml two times a day as needed
  Other Names: Base cream
  Arms: Placebo cream

SUMMARY:
The purpose of this study is to determine if an herbal over-the-counter cream can decrease skin site reactions in multiple sclerosis patients who currently take either Betaseron, Copaxone or Rebif as their subcutaneous medication for managing their multiple sclerosis. Injection site reactions have been indicated as one of the major reasons for discontinuing treatment with the subcutaneous medications (Betaseron, Copaxone, and Rebif) for multiple sclerosis.

DETAILED DESCRIPTION:
Skin site reactions account for one of the most likely reasons for discontinuation of subcutaneous injections of MS medications. It is imperative that additional methods be determined to decrease the reactions and/or treat the reactions that occur. Individuals continue to use over the counter preparations (e.g. Benadryl or steroid creams) or other treatments recently described (warm compresses) to improve tolerance to the subcutaneous injections and the reactions. Both short (3 to 6 months) and long term skin reactions have been reported by patients. They complain about this at office visits and calls to nurses in clinics or to those who teach injection technique. Recently, this investigator and a nurse colleague found that an herbal cream (Bach's Rescue Remedy Cream) reduced the redness and skin site reactions. A small investigator funded mini-pilot demonstrated a decrease in resolution and in size of skin site reactions and satisfaction of herbal cream versus the placebo cream. This proposed research study builds upon Moore's previous success that documented significant decrease in injection site reactions by adding an air bubble to the injection before injection, which is now described in the injection instructions of Copaxone, Rebif, and Axonex. The specific hypotheses for this study as end points include:

1. The herbal cream will significantly decrease time of redness based on daily measure of skin site reactions compared to placebo cream.
2. The herbal cream will decrease discomfort of skin site reactions as measured by a visual analogue scale compared to the placebo cream.
3. Participants will indicate how the herbal cream has made a difference to their quality of life based on a qualitative description of effects of skin site reactions before herbal cream and following use of herbal cream

ELIGIBILITY:
Inclusion Criteria:

* Participants must demonstrate redness of skin site reactions
* Must demonstrate accurate injection technique prior to initiating the study

Exclusion Criteria:

* Cannot read the flexible measure and record the results.
* Are diagnosed with secondary progressive, primary progressive or Devic's MS.
* Are not taking one of the three subcutaneous injections (Betaseron®, Copaxone® or Rebif®).
* Are pregnant.
* Are younger than 18 years of age.
* Are using combination therapy (e.g., 2 of the immunomodulators, chemotherapy)
* Have allergies to any topical creams used on skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Significant decrease in time and size of redness based on daily measure of skin site reactions using herbal cream compared to placebo cream. | 7 days from each injection

SECONDARY OUTCOMES:
Participants will indicate how the herbal cream has made a difference to their quality of life based on a qualitative description of effects of skin site reactions before herbal cream and following use of herbal cream | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Moore, EdD, APRN, Principal Investigator — University of North Carolina at Charlotte
Locations (1):
- University of North Carolina at Charlotte, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Gaines AR, Varricchio F. Interferon beta-1b injection site reactions and necroses. Mult Scler. 1998 Apr;4(2):70-3. doi: 10.1177/135245859800400205. PMID 9599336
- [Background] Moore LA, Kaufman MD, Algozzine R, Irish N, Martin M, Posey CR. Adherence to therapy: using an evidence-based protocol. Rehabil Nurs. 2007 Nov-Dec;32(6):227-32. doi: 10.1002/j.2048-7940.2007.tb00179.x. PMID 18065143
- [Background] Halper J, Harris C, Machler B. Manageing injection-site reactions in patients with MS. Multiple Sclerosis Counseling Points 1:1-10,2005
- [Background] Jolly H, Simpson K, Bishop B, Hunter H, Newell C, Denney D, Oleen-Burkey M. Impact of warm compresses on local injection-site reactions with self-administered glatiramer acetate. J Neurosci Nurs. 2008 Aug;40(4):232-9. doi: 10.1097/01376517-200808000-00007. PMID 18727339
- [Background] Samuel L, Lowenstein EJ. Recurrent injection site reactions from interferon beta 1-b. J Drugs Dermatol. 2006 Apr;5(4):366-7. PMID 16673806